CLINICAL TRIAL: NCT07202975
Title: RE-SCALE: Rehabilitation Engagement and Scaled Access With eXtended Reality and Artificial Intelligence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Hospital Vall d'Hebron (Other); Villa Beretta Rehabilitation Research innovation Institute (Unknown); German Research Center for Artificial Intelligence (DFKI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE-SCALE
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP)

STUDY DESIGN:
Intervention Model Description: Two-site randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed realities rehabilitation program (Experimental): 1. Two sessions at the hospital: one session with traditional exercise + one session with traditional exercise and training with XR system ( 2 weeks)
  2. Four more sessions at home with therapist (L1 therapist and L1 patients) (4 weeks)
  3. Former sessions (until 120 days) with L3 therapist and L1 and L3 patients.
  Interventions: Other: Mixed realities rehabilitation program
- Usual Care (Active Comparator): Group rehabilitation sessions: 8 weeks
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Mixed realities rehabilitation program — 1. Two sessions at the hospital: one session with traditional exercise + one session with traditional exercise and training with XR system ( 2 weeks)
  2. Four more sessions at home with therapist (L1 therapist and L1 patients) (4 weeks)
  3. Former sessions (until 120 days) with L3 therapist and L1 and L3 patients. Usual care: Group rehabilitation sessions: 8 weeks
  Arms: Mixed realities rehabilitation program
Other: Usual Care — Group rehabilitation sessions: 8 weeks
  Arms: Usual Care

SUMMARY:
Background Chronic musculoskeletal pain, especially chronic low back pain (CLBP), is the leading cause of disability worldwide, with a burden expected to rise due to aging and increased longevity. Despite strong evidence supporting multimodal and non-pharmacological management-particularly active physical therapy and self-management-clinical practice still shows low adherence to guidelines, with excessive reliance on imaging, rest, injections, and surgery.

Adherence to physical therapy remains one of the most significant barriers: only 40-50% of patients follow prescribed exercise programs. Factors include kinesiophobia, low motivation, and logistical obstacles. Mixed realities (XR: VR, AR, MR) offer solutions by enhancing motivation, reducing barriers, and personalizing rehabilitation. Evidence from systematic reviews shows VR-based rehabilitation can reduce pain, disability, and kinesiophobia, with immersive VR offering additional benefits like presence and habit-building.

The SHARESPACE project developed and tested a novel XR rehabilitation environment for CLBP that integrates immersive VR/AR, tele-rehabilitation, real-time motor tracking, avatars for social support, and cognitive architectures for synchronization. Usability studies with patients, clinicians, and the general population confirm its feasibility and acceptance. SHARESPACE has completed phases 1 and 2 of XR intervention development (design and feasibility), now aiming to move to phase 3: large-scale clinical validation.

Objectives The main goal is to evaluate not only short-term efficacy but long-term, as well as including more accurate and objective measures. A second objective is the commercial exploitation WE will valuate the efficacy, adherence, and cost-effectiveness of the SHARESPACE XR rehabilitation system compared to usual care in patients with CLBP.

Specific objectives include:

1. To conduct a two-site randomized controlled trial (RCT) comparing XR rehabilitation with conventional group rehabilitation.
2. To assess both short-term and long-term outcomes (pain intensity, disability, kinesiophobia).
3. To monitor and improve adherence through ecological momentary assessment and intervention (EMA/EMI) using an app and activity trackers.
4. To enhance motivation and engagement with gamification, social connectedness, and avatar-based interaction.
5. To generate evidence for commercial exploitation and integration into health systems.

Methodology

The project will conduct a two-site RCT with CLBP patients. Participants will be randomly allocated to:

* XR rehabilitation:

  * Two hospital sessions (traditional + XR-assisted training).
  * Four remote XR sessions with therapist and patients (L1 avatars).
  * Continued home-based XR with automated therapist avatars (L3) for up to 120 days.
  * Integration of EMA/EMI via an app and wearable devices to monitor daily activity, sleep, and adherence, with automated prompts to encourage compliance.
* Usual care: standard group rehabilitation sessions for 8 weeks.

Primary outcomes:

* Pain intensity (VAS, BPI).
* Disability (Oswestry Disability Index).
* Kinesiophobia (Tampa Scale of Kinesiophobia). Secondary outcomes: adherence rates, motivation, patient satisfaction, feasibility, and cost-effectiveness. Motor performance data will be captured in real time via XR tracking and transmitted to therapists for feedback.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Adults over 18 and under 70
* Diagnosis of chronic low back pain with or without radiculopathy
* Minimum of moderate disability (21% ODI score)
* Acceptance of participation and signed consent form
* Internet access at home

Exclusion Criteria:

* History of spinal surgery or fracture
* Signs of upper motor neuron injury: bilateral paresthesia, hyperreflexia, or spasticity, or other negative signs such as fractures
* Other severe medical or psychological conditions that prevent participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity by VAS (0-100mm) | Baseline, through study completion, an average of 8 week and follow-up at 6, 12 and 18
  Significant change at 25 mm
Pain intensity by Brief Pain Inventory | Baseline, through study completion, an average of 8 week and follow-up at 6, 12 and 18
Pain disability by Oswestry Disability Index (ODI) | Baseline, through study completion, an average of 8 week and follow-up at 6, 12 and 18
Pain Kinesiophobia by Tampa Scale of Kinesiophobia (TSK) | Baseline, through study completion, an average of 8 week and follow-up at 6, 12 and 18

REFERENCES:
- [Background] Hoffman HG, Fontenot MR, Garcia-Palacios A, Greenleaf WJ, Alhalabi W, Curatolo M, Flor H. Adding tactile feedback increases avatar ownership and makes virtual reality more effective at reducing pain in a randomized crossover study. Sci Rep. 2023 May 22;13(1):7915. doi: 10.1038/s41598-023-31038-4. PMID 37217536
- See also: Related Info — https://sharespace.eu/partners/universitat-jaume-i/